CLINICAL TRIAL: NCT06803004
Title: Blinded Randomized Control Trail of Artificial Intelligence-Assisted Ultrasound Screening for Neonatal Hip Dysplasia in a Clinical Cohort
Brief Title: Diagnostic Efficacy Study of AI System in Screening Infants With Developmental Dysplasia of the Hip
Acronym: ASIDDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Lixin Jiang, Director of Department of ultrasound in medicine, Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LY2025-004-C
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hip Dysplasia, Developmental
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Junior Sonographer Annotation (Active Comparator): Participants will not receive visual cues from the DeepDDH system. Junior sonographer technicians will offer preliminary interpretations before these are subjected to validation and subsequent review by expert's team.
  Interventions: Other: Junior sonographer measurement of DDH
- Senior Sonographer Annotation (Active Comparator): Participants will not receive visual cues from the DeepDDH system. Senior sonographer technicians will offer preliminary interpretations before these are subjected to validation and subsequent review by expert's team.
  Interventions: Other: Senior sonographer measurement of DDH
- DeepDDH system Annotation (Experimental): Through randomization, a subset of the preliminary interpretations will be conducted by AI technology, and the study team will evaluate the degree of divergence between these AI-generated preliminary interpretations and the final interpretations.
  Interventions: Other: Automated annotation of the DDH measurement through deep learning
- DeepDDH-assist Junior Sonographer Annotation (Experimental): Participants will receive visual cues from the DeepDDH system.
  Interventions: Other: AI-assisted junior sonographer measurement of DDH

INTERVENTIONS:
Other: Junior sonographer measurement of DDH — Participants will not receive visual cues from the DeepDDH system. Junior sonographer technicians will offer preliminary interpretations before these are subjected to validation and subsequent review by expert's team.
  Arms: Junior Sonographer Annotation
Other: Senior sonographer measurement of DDH — Participants will not receive visual cues from the DeepDDH system. Senior sonographer technicians will offer preliminary interpretations before these are subjected to validation and subsequent review by expert's team.
  Arms: Senior Sonographer Annotation
Other: Automated annotation of the DDH measurement through deep learning — Through randomization, a subset of the preliminary interpretations will be conducted by AI technology, and the study team will evaluate the degree of divergence between these AI-generated preliminary interpretations and the final interpretations.
  Arms: DeepDDH system Annotation
Other: AI-assisted junior sonographer measurement of DDH — Participants will receive visual cues from the DeepDDH system.
  Arms: DeepDDH-assist Junior Sonographer Annotation

SUMMARY:
To ascertain the efficacy of the DeepDDH system, a deep learning framework, in enhancing diagnostic accuracy and curtailing follow-up intervals for infants undergoing screening for developmental dysplasia of the hip (DDH), the researchers are executing a blinded, randomized controlled trial. This trial juxtaposes AI-only and AI-assisted assessments of DDH against sonographer interpretations across various proficiency levels in the preliminary analysis of ultrasound images.

DETAILED DESCRIPTION:
1. Participating centers and doctors:

   The data in the ultrasound screening sequence database in this part of the study were mainly from Renji Hospital and the Sixth People's Hospital in Shanghai between August 2014 and December 2021. Renji Hospital, the Sixth People's Hospital, and the Pediatric Hospital Affiliated to Fudan University, three top-three hospitals in Shanghai, started Graf ultrasound examination earlier, with an average history of more than 10 years. And they are responsible for providing expert sonographers with more than 5-10 years of DDH ultrasound diagnosis experience, and pediatric orthopedic experts with 5-10 years of DDH diagnosis experience to participate in the study. However, several other primary or remote medical institutions with late DDH ultrasound screening and insufficient diagnostic experience were mainly responsible for providing primary sonographers to participate in the study. Before the study, the sonographers involved in this study will be evaluated uniformly and quantitatively through examination papers.
2. Research process:

One week before the start of the study, the sonographers registered in the study received uniform training of the latest DDH ultrasound diagnosis in the form of PPT, video, literature study, and offline instruction.

For the included cases in the ultrasound screening sequence database, they would appear in different control groups in a random form, such as the AI model, the Expert sonographer group, the primary sonographer group, and the primary sonographer with AI 'aid group. All cases in the ultrasound screening sequence database were stratified and block-randomized into the above four groups (primary, experts, AI-independent, AI-assisted primary).

In the AI-assisted group, each sonographer was asked to choose whether to modify or confirm the diagnosis according to the measurement marks, diagnostic angles and typing results provided by the AI device. However, in the Expert sonographer group and junior sonographer unassisted group, the dedicated research assistant will turn off the AI display function to ensure that no additional information is provided to the sonographer. The consensus of two pediatric orthopedic expert with 5-10 years of experience in DDH ultrasound diagnosis was used as the gold standard. In case of disagreement, a third pediatric expert will evaluate the diagnosis results of DDH. The final consensus was used as the gold standard.

Then, the pediatric orthopedic expert group were given the initial annotations diagnosis results of DDH in the above four groups, including diagnostic images, diagnostic measurement marks, diagnostic angles and diagnostic types. And by reviewing the initial annotations, selecting "confirm" or "modify" the initial annotations, the final annotations are made again for those who need to be modified, and the final report results are obtained.

Finally, the operation results of the above different groups were summarized and analyzed by independent research assistants, including α Angle, β Angle, typing results, and the specific follow-up experience of the case including follow-up times, diagnosis time, Bang's index, proportion of studies the annotation is changed, proportion of studies the DDH type is changed in final report, and mean change in alpha angle between preliminary and final report.

ELIGIBILITY:
Inclusion Criteria:

* Infants underwent DDH ultrasound examinations.
* Infants aged 28 days to 6 months.

Exclusion Criteria:

* Infants with lacking or incomplete ultrasound images.
* Infants with poor image quality, including non-compliance with anatomical identification and usability check.
* Infants with hip dysplasia caused by other diseases.

Ages: 28 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1789 (Actual)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Average diagnostic accuracy | up to 4 weeks
  It is calculated by dividing the number of preliminary interpretations that are consistent with the expert team's grading by the total number of cases that should be diagnosed.

SECONDARY OUTCOMES:
Average diagnostic sensitivity | up to 4 weeks
  It is calculated by dividing the number of true positive cases by the sum of true positive cases and false negative cases.
Average diagnostic specificity | up to 4 weeks
  It is calculated by dividing the number of true negative cases by the sum of true negative cases and false positive cases.
Average times of follow-up visits | up to 4 weeks
  The average number of follow-up visits for each group is obtained by dividing the total number of follow-up visits for each participating infant within the group by the number of participating infants in that group.
Diagnosis time | up to 4 weeks
  Time taken to make ultrasound diagnosis in each group
Bang's index | up to 4 weeks
  Bang's index is used to evaluate whether the blind method is implemented successfully
Frequency pediatrician adjusts preliminary annotation | up to 4 weeks
  Proportion of studies the annotation is changed
Frequency pediatrician adjusts preliminary DDH type | up to 4 weeks
  Proportion of studies the DDH type is changed in final report
Mean change in alpha angle between preliminary and final report | up to 4 weeks
  Average change in alpha angle between preliminary and final report

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical demographic information of the subjects was recorded through the Case Record Form, and the data will be collected and managed electronically through the ResMan platform.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code